CLINICAL TRIAL: NCT07111182
Title: ATM 5-ALA: Intraoperative Fluorescence-Guided Aspirate Tissue Monitoring of 5-ALA During Brain Tumor Surgery
Brief Title: Intraoperative Fluorescence-Guided Aspirate Tissue Monitoring of 5-ALA During Brain Tumor Surgery
Acronym: ATM5-ALA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Marginum Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2025-0505
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: In general, the current literature favors more and more aggressive treatments for high-grade III-IV (Barak et al. 2021), grade II (Rossi et al. 2020), and both non-symptomatic and symptomatic low-grade gliomas with progressive features (Zeng et al. 2021).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Usability Assessment (Other): Neurosurgeons and surgical nurses have assessed the usability, performance and safety of the device based on operation video recordings or user testing with high-grade glioma-simulating synthetic phantoms.
  neurosurgeons will use the HIVEN® during high-grade glioma surgeries in patients in authentic conditions according to the intended use and IFU and assessed its performance and benefit-risk profile. Surgical nurses gave feedback on the device's preoperative preparations and usability during the interventional study.
  Interventions: Device: HIVEN Medical Device

INTERVENTIONS:
Device: HIVEN Medical Device — A medical device (HIVEN®) detects 5-ALA-induced fluorescence from the surgical suction and gives sound feedback to the operating surgeon indicating tumor tissue and overcoming the challenges is the contemporary FGS methods. The device is used for detecting fluorescence of flowing tissues within a transparent tube and providing auditory feedback of tissue fluorescence for neurosurgeons. There is no patient contact intended with this device.

SUMMARY:
Gliomas are tumors that occur in all ages; they include the most common malign primary central nervous system tumors in developed countries. Gliomas are often aggressive, and their recommended treatment is surgical resection and chemoradiation. Complete tumor removal is challenging because of diffuse cell growth and the proximity of functionally critical tissues. The current golden standard for intraoperative glioma detection is fluorescence-guided surgery (FGS) using 5-ALA. In 5-ALA FGS the drug-induced fluorescence helps to visually detect tumor cells, which improves resection rates and delays tumor progression. Tumor cells are often left unnoticed because of visual obstacles or weak fluorescence, which may lead to local recurrence and reoperations. Surgical suction devices are routinely used to remove cancerous tissues, but so far, the analysis of the suction waste has not been used in near real-time tissue detection.

DETAILED DESCRIPTION:
A novel medical device (HIVEN®) detects 5-ALA-induced fluorescence from the surgical suction and gives sound feedback to the operating surgeon indicating tumor tissue and overcoming the challenges is the contemporary FGS methods. The 5-ALA (Gleolan, NX Development Corp) has been already FDA-approved since 2017 for fluorescence-guided resection of suspected WHO grade 3 or 4 gliomas. The HIVEN® device has been investigated in Europe during 33 surgeries and the MDR (EU) 2017/745 approval was granted on 09/2025.The device is commercially available in the EU starting from 09/2025. The CE mark is approved for a Class IIb device risk classification. The current medical device study aims to demonstrate the feasibility and the benefit-risk ratio of HIVEN® for detecting tumor fluorescence from the surgical suction waste as a part of the FDA medical device process. The feedback from the device is expected to provide supplementary information on fluorescence and add value to fluorescence-guided surgical workflow.

ELIGIBILITY:
Inclusion Criteria:-

* Patient admitted to neurosurgery department for surgical resection of a suspected grade 3 or 4 glioma with 5-ALA (cases)
* Patient admitted to neurosurgery department for surgical resection of a primary of secondary brain tumor with no 5-ALA (controls)
* Patients aged 18 years old or older (all patients)
* Informed consent obtained (all patients)

Exclusion Criteria:

* Patient belongs to the following vulnerable groups: children, pregnant, prisoners or intellectually disabled.
* The participants are not randomized. Randomization is not conducted as the number of eligible patients is limited, subjecting to a long recruitment period that reciprocally increases the bias from uncontrollable (evolving) surgical techniques and adjunct treatments.
* The patients are screened and informed of the study before the surgical operation and enrolled after verification of eligibility and written informed consent has been received.

Potential study participants are identified from the clinic's planned or urgent surgeries list. The participants are contacted before the operation by the research staff and/or the physician responsible for the treatment. The participants are provided with written and oral information about the research and the time to consider their participation. Finally, the participants are asked for their informed consent and enrolled to the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the increased detection of fluorescence during surgery (performance) | During procedure video recording
  Fluorescence detection rate during surgery measured per seconds of video (performance)
Assess the safety and benefit-risk profile versus a legally marketed alternative therapy i.e. visual fluorescence guidance (safety) | During procedure user's questionnaires
  Benefit-risk profile based on user's systematic questionnaires indicates non-inferiority to visual fluorescence guidance (safety)

CONTACTS AND LOCATIONS:
Overall Officials: Fady T Charbel, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States